CLINICAL TRIAL: NCT03236168
Title: Impact of Community Scabies Treatment on Head Lice Prevalence in the Solomon Islands
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14257
Record Dates: First submitted 2017-07-26; First posted 2017-08-01 (Actual); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-11

CONDITIONS: Scabies; Head Lice
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): This study consists of a single treatment arm. Patients will receive Ivermectin or where contraindicated (Pregnancy, Breastfeeding, Weight <15kg) Permethrin Cream and Malathion shampoo
  Interventions: Drug: Ivermectin; Drug: Permethrin 5%; Drug: Malathion Shampoo 0.5%

INTERVENTIONS:
Drug: Ivermectin — A single weight based dose of ivermectin
Drug: Permethrin 5% — Permethrin cream is used in conjunction with Malathion shampoo when ivermectin is contra-indicated
Drug: Malathion Shampoo 0.5% — Permethrin cream is used in conjunction with Malathion shampoo when ivermectin is contra-indicated

SUMMARY:
This is a pilot study evaluating if treatment for scabies also treats headlice in the same community

DETAILED DESCRIPTION:
Background:

Scabies and head lice are both ubiquitous ectoparasitic infections that have been identified as common public health problems in the Pacific Island Country Territories. Mass drug administration using ivermectin is increasingly recognised as an effective strategy for scabies treatment and control, however, its possible impact on prevalence of head lice has not been evaluated. Given that oral ivermectin is an effective treatment option for pediculosis capitis, we hypothesise that community treatment with ivermectin for scabies would also provide benefit by reducing prevalence of head lice infestation in the community. We aim to test this hypothesis with a small-scale pilot study in the Solomon Islands.

Methodology:

The study would be carried out at the Atoifi Adventist Hospital campus, on the North-Eastern coast of the island of Malaita. The campus houses an estimated 180 individuals and all residents would be invited to participate in the study and be offered treatment.

At baseline all individuals would undergo a standardized examination to collect data on the presence of scabies, impetigo and head lice. Following examination individuals would be weighed and given directly observed standard treatment for scabies.

Treatment for scabies consists of one oral dose of ivermectin (200 micrograms per kilogram) at day 1 and at day 8.

Individuals with contra-indications (pregnancy, breast feeding, weight under 15kg) would be offered the alternative of 5% permethrin cream and malathion shampoo.

Individuals would be re-examined at 48hours (to assess immediate killing of head lice) and again at 2 weeks. Final follow-up will be at 3 months to establish: 1) whether changes in head lice prevalence have been sustained 2) what the impact of treatment on scabies and impetigo with ivermectin is in this specific community.

ELIGIBILITY:
Inclusion Criteria:

* All participants living in the community will be offered treatment

Exclusion Criteria:

* Patients with a contradindication to study medication
* Patients unable to provide consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atoifi Adventist Hospital, Atoifi, Malaita Province, Solomon Islands

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be made available alongside any future publications

REFERENCES:
- [Derived] Coscione S, Esau T, Kekeubata E, Diau J, Asugeni R, MacLaren D, Steer AC, Kositz C, Marks M. Impact of ivermectin administered for scabies treatment on the prevalence of head lice in Atoifi, Solomon Islands. PLoS Negl Trop Dis. 2018 Sep 25;12(9):e0006825. doi: 10.1371/journal.pntd.0006825. eCollection 2018 Sep. PMID 30252856

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 118
Completed | 107
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 118
Age, Customized [Count of Participants; unit: Participants]
  <= 10 years | 32
  11-20 years | 31
  >= 21 years | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 118
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Solomon Islands | 118
Headline Prevalence [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Headlice
Description: Assessed in the study population by physical examination of hair
Time Frame: 2 Weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 117
Participants | 3

2. Secondary Outcome: Number of Participants With Headlice
Description: Assessed in the study population by physical examination of hair
Time Frame: 48hrs after treatment
Reporting Status: Not Posted

3. Secondary Outcome: Number of Participants With Headlice
Description: Assessed in the study population by physical examination of hair
Time Frame: 3 Months after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03236168/Prot_SAP_000.pdf